CLINICAL TRIAL: NCT03888911
Title: Double-blind, Randomized, Three-armed, Placebo-controlled, Clinical Investigation to Evaluate the Benefit and Tolerability of Two Dosages of IQP-LU-104 in Reducing Body Weight in Overweight and Moderately Obese Subjects
Brief Title: Benefit and Tolerability of IQP-LU-104 in Weight Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: InQpharm Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: INQ/011618
Record Dates: First submitted 2019-03-20; First posted 2019-03-25 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Overweight; Obesity
Keywords: Flaxseed mucilage; Weight loss; Satiety
MeSH Terms: conditions — Overweight; Obesity; Weight Loss

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High dose IQP-LU-104 (5120mg) (Experimental): High dose treatment group
  Interventions: Dietary Supplement: High dose IQP-LU-104 (5120mg)
- Low dose IQP-LU-104 (2560mg) (Experimental): Low dose treatment group
  Interventions: Dietary Supplement: Low dose IQP-LU-104 (2560mg)
- Placebo (Placebo Comparator): Placebo group
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: High dose IQP-LU-104 (5120mg) — 1 sachet to be taken 2 times daily orally, together with 2 main meals
  Arms: High dose IQP-LU-104 (5120mg)
Dietary Supplement: Low dose IQP-LU-104 (2560mg) — 1 sachet to be taken 2 times daily orally, together with 2 main meals
  Arms: Low dose IQP-LU-104 (2560mg)
Dietary Supplement: Placebo — 1 sachet to be taken 2 times daily orally, together with 2 main meals
  Arms: Placebo

SUMMARY:
This study is to evaluate the benefit and tolerability of two dosages of IQP-LU-104 (5120mg and 2560mg daily) in reducing body weight in overweight and moderately obese subjects

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 65 years
2. Overweight (BMI 25 to < 30 kg/m2) and moderately obese (BMI 30 to < 35 kg/m2) subjects
3. Generally in good health
4. Desire to lose weight
5. Accustomed to regular daily consumption of 3 main meals (breakfast, lunch, dinner)
6. Consistent and stable body weight in the last 3 months prior to V1 (less than 5% self-reported change)
7. Subject's agreement to comply with study procedures, in particular:

   * to take IP as recommended
   * to follow diet recommendation during the study
   * to complete the subject diary and study questionnaires
   * to maintain the habitual level of physical activity during the study
8. Women of childbearing potential:

   * commitment to use contraception methods
   * negative pregnancy testing (beta human chorionic gonadotropin test in urine) at V1
9. Consents to participate, understands requirements of the study and is willing to comply

Exclusion Criteria:

1. Known sensitivity to the ingredients of the investigational product or source of ingredients
2. History and/or presence of clinically significant condition/disorder, which per investigator's judgment could interfere with the results of the study or the safety of the subject, e.g.:

   * untreated or non-stabilised thyroid gland disorder
   * untreated or non-stabilised hypertension (regular systolic blood pressure ≥ 140 mmHg and/or diastolic blood pressure ≥ 90 mmHg)
   * acute or chronic gastrointestinal (GI) disease or digestion/absorption disorders (e.g. inflammatory bowel disease, coeliac disease, pancreatitis etc.)
   * diabetes mellitus type 1
   * untreated or non-stabilised diabetes mellitus type 2
   * any other relevant serious organ or systemic diseases
3. Significant surgery within the last 6 months prior to V1:

   * GI surgery
   * liposuction
4. History of eating disorders like bulimia, anorexia nervosa, binge-eating within the last 12 months prior to V1
5. Deviation of safety laboratory parameter(s) at V1 that is:

   * clinically significant or
   * > 2x upper limit of normal, unless the deviation is justified by a previously known not clinically relevant condition (e.g. Gilbert's syndrome)
6. Any electronic medical implant
7. Regular medication and/or supplementation and/or treatment within the last month prior to V1 and during the study, which per investigator's judgment could interfere with the results of the study or the safety of the subject, e.g.:

   * that could influence body weight (e.g. systemic cortcosteroids, antipsychotics, anti-depressants)
   * that could influence gastrointestinal functions (e.g. antibiotics, laxatives, opioids, anticholinergics etc.) as per investigator judgment
   * for weight management (e.g. fat binder, carbohydrate/starch blocker, fat burner, satiety products etc.)
   * any other relevant medication and/or supplementation
8. Diet/weight loss programs within the last 3 months prior to V1 and during the study
9. Smoking cessation within 6 months prior to V1 or during the study (regular smoking during the study at the same level as prior to the study is allowed)
10. Vegetarian, vegan or other restrictive diet
11. Women of child-bearing potential: pregnancy or nursing
12. History of or current abuse of drugs, alcohol or medication
13. Participation in another clinical study in the 30 days prior to V1 and during the study
14. Any other reason for exclusion as per investigator's judgment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2019-03-05 (Actual); Primary Completion 2019-11-21 (Actual); Study Completion 2019-11-21 (Actual)

PRIMARY OUTCOMES:
Mean change in body weight (kg) | 12 weeks
  Difference in mean change of body weight (kg) between the higher dosed verum and placebo group after 12 weeks of intervention in comparison to baseline
Mean change in body weight (kg) | 12 weeks
  Difference in mean change of body weight (kg) between the lower dosed verum and placebo group after 12 weeks of intervention in comparison to baseline

SECONDARY OUTCOMES:
Mean change in body weight (kg) | 4 and 8 weeks
  Difference between the higher dosed verum and placebo group in mean change of body weight (kg) after 4 and 8 weeks of intervention, each in comparison to baseline
Mean change in body weight (kg) | 4 and 8 weeks
  Difference between the lower dosed verum and placebo group in mean change of body weight (kg) after 4 and 8 weeks of intervention, each in comparison to baseline
Body weight (kg) | 4, 8, 12 weeks
  Difference between the two verum and placebo groups in body weight (kg) after 4, 8, and 12 weeks of intervention
Change in body weight percentage (%) | 4, 8, 12 weeks
  Difference between the two verum and placebo groups in the changes in body weight (%) after 4, 8, and 12 weeks of intervention, each in comparison to baseline
Proportion of subjects with weight loss | 4, 8, 12 weeks
  Difference between the two verum and placebo groups in the proportion of subjects who lost at least 3%, 5% and 10% of baseline body weight after 4, 8, and 12 weeks of intervention, each in comparison to baseline
Waist circumference (cm) | 4, 8, 12 weeks
  Difference between the two verum and placebo groups in waist circumference (cm) after 4, 8, and 12 weeks of intervention
Change in waist circumference (cm) | 4, 8, 12 weeks
  Difference between the two verum and placebo groups in the changes in waist circumference (cm) after 4, 8, and 12 weeks of intervention, each in comparison to baseline
Hip circumference (cm) | 4, 8, 12 weeks
  Difference between the two verum and placebo groups in hip circumference (cm) after 4, 8, and 12 weeks of intervention
Change in hip circumference (cm) | 4, 8, 12 weeks
  Difference between the two verum and placebo groups in the changes in hip circumference (cm) after 4, 8, and 12 weeks of intervention, each in comparison to baseline
Waist-hip ratio | 4, 8, 12 weeks
  Difference between the two verum and placebo groups in waist-hip ratio after 4, 8, and 12 weeks of intervention
Change in waist-hip ratio | 4, 8, 12 weeks
  Difference between the two verum and placebo groups in the changes in waist-hip ratio after 4, 8, and 12 weeks of intervention, each in comparison to baseline
BMI (kg/m^2) | 4, 8, 12 weeks
  Difference between the two verum and placebo groups in BMI (kg/m^2) after 4, 8, and 12 weeks of intervention
Change in BMI (kg/m^2) | 4, 8, 12 weeks
  Difference between the two verum and placebo group in the changes in BMI (kg/m^2) after 4, 8, and 12 weeks of intervention, each in comparison to baseline
Body fat percentage (%) | 4, 8, 12 weeks
  Difference between the two verum and placebo groups in body fat (%) after 4, 8, and 12 weeks of intervention
Change in body fat percentage (%) | 4, 8, 12 weeks
  Difference between the two verum and placebo groups in the changes in body fat (%) after 4, 8, and 12 weeks of intervention, each in comparison to baseline
Body fat mass (kg) | 4, 8, 12 weeks
  Difference between the two verum and placebo groups in body fat mass (kg) after 4, 8, and 12 weeks of intervention
Change in body fat mass (kg) | 4, 8, 12 weeks
  Difference between the two verum and placebo groups in the changes in body fat mass (kg) after 4, 8, and 12 weeks of intervention, each in comparison to baseline
Fat free mass (kg) | 4, 8, 12 weeks
  Difference between the two verum and placebo groups in fat free mass (kg) after 4, 8, and 12 weeks of intervention
Change in fat free mass (kg) | 4, 8, 12 weeks
  Difference between the two verum and placebo groups in the changes in fat free mass (kg) after 4, 8, and 12 weeks of intervention, each in comparison to baseline
Evaluation of feeling of hunger using visual analogue scales (VAS) | 4, 8, 12 weeks
  Difference between the two verum and placebo groups in the evaluation of feelings of hunger using VAS after 4, 8, and 12 weeks of intervention
Change in the evaluation of feeling of hunger using visual analogue scales (VAS) | 4, 8, 12 weeks
  Difference between the two verum and placebo groups in the changes in evaluation of feelings of hunger using VAS after 4, 8, and 12 weeks of intervention, each in comparison to baseline
Evaluation of feeling of satiety using visual analogue scales (VAS) | 4, 8, 12 weeks
  Difference between the two verum and placebo groups in the evaluation of feelings of satiety using VAS after 4, 8, and 12 weeks of intervention
Change in the evaluation of feeling of satiety using visual analogue scales (VAS) | 4, 8, 12 weeks
  Difference between the two verum and placebo groups in the changes in evaluation of feelings of satiety using VAS after 4, 8, and 12 weeks of intervention, each in comparison to baseline
Evaluation of feeling of fullness using visual analogue scales (VAS) | 4, 8, 12 weeks
  Difference between the two verum and placebo groups in the evaluation of feelings of fullness using VAS after 4, 8, and 12 weeks of intervention
Change in the evaluation of feeling of fullness using visual analogue scales (VAS) | 4, 8, 12 weeks
  Difference between the two verum and placebo groups in the changes in evaluation of feelings of fullness using VAS after 4, 8, and 12 weeks of intervention, each in comparison to baseline
Evaluation of feeling of craving using visual analogue scales (VAS) | 4, 8, 12 weeks
  Difference between the two verum and placebo groups in the evaluation of feelings of craving using VAS after 4, 8, and 12 weeks of intervention
Change in the evaluation of feeling of craving using visual analogue scales (VAS) | 4, 8, 12 weeks
  Difference between the two verum and placebo groups in the changes in evaluation of feelings of craving using VAS after 4, 8, and 12 weeks of intervention, each in comparison to baseline
Change in the quality of life using Impact of Weight on Quality of Life (IWQOL-Lite) Questionnaire | 4, 8, 12 weeks
  Difference between the two verum and placebo groups in the changes in quality of life using (IWQOL-Lite) questionnaire after 4, 8 and 12 weeks of intervention, each in comparison to baseline
Lipid metabolism parameters (mmol/l) | 12 weeks
  Difference between the two verum and placebo groups in total cholesterol (mmol/l), LDL-cholesterol (mmol) and HDL cholesterol (mmol) after 12 weeks of intervention
Change in lipid metabolism parameters (mmol/l) | 12 weeks
  Difference between the two verum and placebo groups in the changes in lipid metabolism parameters after 12 weeks of intervention, each in comparison to baseline
HbA1C percentage (%) | 12 weeks
  Difference between the two verum and placebo groups in HbA1C (%) after 12 weeks of intervention
Change in HbA1C percentage (%) | 12 weeks
  Difference between the two verum and placebo groups in the changes in HbA1C (%) after 12 weeks of intervention, each in comparison to baseline

OTHER OUTCOMES:
Safety parameters (lab parameters and vital signs) | 12 weeks
  Assessment of laboratory results in full blood count, clinical chemistry, blood pressure and pulse rate

CONTACTS AND LOCATIONS:
Overall Officials: Udo Bongartz, MD, PhD, Principal Investigator — Analyze & Realize
Locations (1):
- Analyze & Realize, Berlin, Germany

REFERENCES:
- [Derived] Bongartz U, Hochmann U, Grube B, Uebelhack R, Alt F, Erlenbeck C, Peng LV, Chong PW, De Costa P. Flaxseed Mucilage (IQP-LU-104) Reduces Body Weight in Overweight and Moderately Obese Individuals in a 12-week, Three-Arm, Double-Blind, Randomized, and Placebo-Controlled Clinical Study. Obes Facts. 2022;15(3):395-404. doi: 10.1159/000522082. Epub 2022 Feb 7. PMID 35130547